CLINICAL TRIAL: NCT04174183
Title: Evaluation of the Effectiveness of a Closed-incision Negative-pressure Therapy (Prevena®) on Bilateral Groin Incision
Acronym: PREVISION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A02416-51
Record Dates: First submitted 2019-11-14; First posted 2019-11-22 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2019-10

CONDITIONS: Bilateral Vascular Groin Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevena (right side) - Dry dressing (left side) (Experimental)
  Interventions: Device: Closed-incision Negative-pressure Therapy - Dry dressing
- Prevena (left side) - Dry dressing (right side) (Experimental)
  Interventions: Device: Closed-incision Negative-pressure Therapy - Dry dressing

INTERVENTIONS:
Device: Closed-incision Negative-pressure Therapy - Dry dressing — A Closed-incision Negative-pressure Therapy is applied on one groin incision - A dry dressing is applied on one groin incision .

SUMMARY:
Closed-incision negative-pressure therapy are medical device that are suspected to reduce groin wound complication in vascular surgery. The aim of this study is to compareon on the same patient a Closed-incision negative-pressure therapy (Prevena®, KCI) versus a traditional gauze dressings after a bilateral vascular groin surgery. To do this, each device is applied on one groin incision and the side, left or right, is randomized.

DETAILED DESCRIPTION:
The prevalence of surgical site infections in groin vascular surgery is 3-44%. The factors causing these infections are well identified: disruption of lymphatic vessels, proximity of genital organs, presence of prosthetic material, etc. The risk of developing an infection of the surgical site is also influenced by the patient's comorbidities and by the surgical context.

Closed-incision negative-pressure therapy are medical device that are suspected to reduce groin wound complication in vascular surgery. The mechanisms of action for negative-pressure therapy include protecting the wound bed, splinting soft tissue, reducing oedema,increasing perfusion and enhancing development of granulation tissue.

Presently, there are no guidelines for the use of this device or not in groin incision and this decision is left to the surgeon's discretion.

The main objective is to demonstrate the superiority of closed-incision negative-pressure therapy over the application of a traditional gauze dressings to reduce the rate of major complications (i.e. requiring an extension of hospitalization time) during bilateral vascular groin surgery. To do this, each device is applied on one groin incision and the side, left or right, is randomized.

The secondary objectives are:

1. To demonstrate the superiority of closed-incision negative-pressure therapy over the application of a dry dressing in reducing the score of complications (major and minor) during vascular groin surgery. The complication score is the number of complications observed during the consultation conducted on day four after the surgery, among the following:

   * Major :

     1. Presence of pus
     2. Bloody and/or lymphatic discharge
     3. Disunity
     4. Necrosis
   * Minor :

     5) Bruising 6) Hematoma 7) Wound extension
2. To compare the rate of major complications between closed-incision negative-pressure therapy and dry dressing application in different clinical settings.

3. To demonstrate the superiority of closed-incision negative-pressure therapy over the application of a dry dressing in reducing the score of complications 2-3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Person affiliated to a health insurance system
* Person who has received full information on the organization of the research and has signed his or her informed consent
* Person presenting a bilateral vascular groin surgery
* Major person

Exclusion Criteria:

* Person with a known allergy to one of the components of the evaluated product (including: acrylic or silver-based adhesives)
* Person with a contraindication to the product(s) being evaluated
* Non-collaborative or agitated patient
* Patients with hemostasis problems
* Persons referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code:
* Pregnant woman, parturient or breastfeeding mother
* Minor person (not emancipated)
* Adult person subject to a legal protection measure (guardianship, curatorship, protection of justice)
* Adult person unable to consent
* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-12-24 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Wound aspect - major complication | 4 days
  Left and right wound incision are inspected and the presence of major complication are reported.
  Major complication :
  Presence of pus Bloody and/or lymphatic discharge Disunity Necrosis

SECONDARY OUTCOMES:
Score of complications | 4-days
  Left and right wound incision are inspected and the presence of major and minor complication are reported. A score of complications is established.
  - Major : Presence of pus Bloody and/or lymphatic discharge Disunity Necrosis
  - Minor : Bruising Hematoma Wound extension
  Each complication amount to 1 point on the complication score.
Major complication in different clinical settings | 4-days
  Left and right wound incision are inspected and the presence of major complication are reported.
  Major complication :
  Presence of pus Bloody and/or lymphatic discharge Disunity Necrosis
  During the analysis, patient are divided into several group depending of the presence or absence of comorbidities.
Wound aspect - major complication (long term) | 2-3 months
  Left and right wound incision are inspected and the presence of major complication are reported.
  Major complication :
  Presence of pus Bloody and/or lymphatic discharge Disunity Necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Nicla Settembre, Principal Investigator — Service de chirurgie vasculaire - Centre Hospitalier Régional Universitaire de Nancy - Allée du Morvan - 54511 Vandœuvre-lès-Nancy Cedex
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Vandœuvre-lès-Nancy, Grand Est, France

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585